CLINICAL TRIAL: NCT06435377
Title: Prospective Observational Study APC AND BIOPSY POST COLD-EMR IN COLONIC LESIONS
Brief Title: Efficacy, Safety and Recurrence After Cold-EMR Plus APC for Large Colonic Lesions
Acronym: EMR+APC
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Cold-EMR plus APC
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Procedure: Cold EMR + APC — * Initial submucosal injection of saline solution and methylene blue, followed by 'piece-meal' resection using a dedicated cold snare
  * Biopsy of the resection bed
  * Ablation of the defect using argon plasma coagulation (APC).

SUMMARY:
This prospective observational study aims to evaluate the efficacy, safety and recurrence of cold-snaring for large colonic lesions combined with argon plasma coagulation of the resection bed.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≧ 18 years undergoing colonoscopy for any indication (screening, anemia, surveillance, or scheduled to undergo endoscopic mucosal resection)
* Lesions of 20 mm and larger.
* All colonic lesions removed using COLD-EMR technique, presenting both adenomatous (Kudo IIIL/IIIS pit pattern)
* Patients who were able to provide written informed consent

Exclusion Criteria:

* Suspected lesions for submucosal invasion (e.g., Kudo V or Paris 0-IIa-IIc with non-granular surface)
* Lesions with a wide Paris 0-Is component (>10mm) that could increase the risk of submucosal invasion and could limit the mechanical cutting of the snare
* Pedunculated polyps
* Active/quiescent colitis
* Rectal lesions
* Residual or recurrent adenoma after endoscopic mucosal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be evaluated for post-procedural pain (using a VAS scale) and need for pain-killers. As part of the standard care, the patient will receive a 30-day post procedure follow-up phone call or an ambulatory evaluation will be arranged 30-days after the endoscopic procedure, to discuss the histologic results and schedule a standard follow-up colonoscopy procedure after the initial procedure. The investigators will measure the post procedural pain in the first four weeks after treatment, the need for pain-killers and, should these occur, the adverse events (included fever, hematochezia, need for hospital admission). The rate of recurrence will be calculated by endoscopic visualization of the EMR site at the follow-up (T1:3-6 months; T2 11-13Months) using endoscopic magnification and electronic chromoendoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Residual | 1 day
  Evaluation of residual in the biopsy of the defect after the cold-EMR. The specimen will be evaluated independently from the polyp sample.
Recurrence | 1 year
  The recurrence rate of adenomas at the site of any qualifying, previously resected lesions is measured after 3-6 and 12 months.

SECONDARY OUTCOMES:
Efficacy of procedure | 1 day
  Complete resection of polyp
Rate of delayed bleeding of the patient | 1 day
  Delayed-bleeding, defined was defined as clinical evidence of bleeding (hematemesis, hematochezia or melena or a decrease of hemoglobin concentration > 2g/dL, which required transfusion or endoscopic reintervention with hemostasis within 30 days of hospital discharge)
Rate of post-polipectomy syndrome | 1 day
  The post-polipectomy syndrome is defined by the presence of fever or abdominal pain
perforation | 1 day
  Rate of perforation and delayed perforation
Time | 1 day
  Average time of procedure and polyp resection time

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided